CLINICAL TRIAL: NCT05896605
Title: Monitoring of Azathioprine Metabolite Concentrations and Cytokine Levels in Neuromyelitis Optica Spectrum Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: First Affiliated Hospital of Guangxi Medical University (Other)
Responsible Party: Principal Investigator, Qingmeng Huang, Mrs., First Affiliated Hospital of Guangxi Medical University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: qingmenghuang
Record Dates: First submitted 2023-05-22; First posted 2023-06-09 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-05

CONDITIONS: NMO Spectrum Disorder; Azathioprine Adverse Reaction
Keywords: NMOSD, AZA, 6-TGN, 6-MMPN, IL-6, NLRP3, IL-18
MeSH Terms: conditions — Neuromyelitis Optica | interventions — Azathioprine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 1 month after AZA treatment (Active Comparator): Before medication, TPMT activity was normal, and azathioprine was started at small doses and added every two weeks after no adverse effects, namely 50 mg qd for two weeks, 50mg bid for two weeks, and maintained at 50mg tid. Low-dose hormone therapy was administered to all patients simultaneously.Blood (5ml) was collected from peripheral veins in 1 month after AZA treatment.
  Interventions: Drug: Azathioprine
- 6 months after AZA treatment (Active Comparator): Before medication, TPMT activity was normal, and azathioprine was started at small doses and added every two weeks after no adverse effects, namely 50 mg qd for two weeks, 50mg bid for two weeks, and maintained at 50mg tid. Low-dose hormone therapy was administered to all patients simultaneously.Blood (5ml) was collected from peripheral veins in 6 months after AZA treatment.
  Interventions: Drug: Azathioprine
- over 1 year after AZA treatment (Active Comparator): Before medication, TPMT activity was normal, and azathioprine was started at small doses and added every two weeks after no adverse effects, namely 50 mg qd for two weeks, 50mg bid for two weeks, and maintained at 50mg tid. Low-dose hormone therapy was administered to all patients simultaneously.Blood (5ml) was collected from peripheral veins over 1 year after AZA treatment.
  Interventions: Drug: Azathioprine
- healthy control (No Intervention): Ten healthy volunteers with physical examination in our hospital were selected as the healthy control (HC) group. Serum samples from healthy controls were collected.

INTERVENTIONS:
Drug: Azathioprine — Before medication, TPMT activity was normal, and AZA was started at small doses and added every two weeks after no AEs, namely 50 mg qd for two weeks, 50mg bid for two weeks, and maintained at 50mg tid.
  Other Names: Azathioprine Tablets
  Arms: 1 month after AZA treatment; 6 months after AZA treatment; over 1 year after AZA treatment

SUMMARY:
Background: The pathogenesis of NMOSD has been linked to the cytokines interleukins (IL) -6, NOD-, LRR-and pyrin domain-containing 3 (NLRP3) and IL-18 that contribute to development of inflammatory reactionsmay. Although azathioprine (AZA) is efficacious in preventing NMOSD recurrence, it may have adverse effects (AEs) maybe related to the plasma concentrations.

Objective: We would monitor the blood concentrations of AZA in NMOSD, and their relationship with cytokines, severity, efficacy, and safety range of the drug.

Methods: A total of 53 NMOSD patients were included in the study, which included 20 patients who had received AZA treatment within 1 month, and 16 patients who had received AZA treatment within 6 months, as well as 17 patients who had received AZA treatment at least 12 months. The patient's immunotherapy regimen was low-dose hormone combined with AZA. AZA was started at small doses and added every two weeks after no AEs, namely 50 mg qd for two weeks, 50mg bid for two weeks, and maintained at 50mg tid. The following clinical data were collected: gender, age, clinical symptoms, EDSS score, number of recurrences and AEs, etc. Healthy controls (HC) comprised 10 individuals. AZA metabolite concentrations 6-thioguaninenucleotides (6-TGN) and 6-methylmercaptopurine nucleotides (6-MMPN) were measured by High-performance liquid chromatography (HPLC). Levels of IL-6, NLRP3 and IL-18 were measured by Enzyme-linked immunosorbent assay (ELISA).

DETAILED DESCRIPTION:
A total of 53 NMOSD patients were recruited from Neurology Department of the First Affiliated Hospital of Guangxi Medical University.According to the duration of AZA treatment, 20 patients were divided into 1 month after AZA treatment, 16 patients in 6 months after AZA treatment and 17 patients over 12 months after AZA treatment. Clinical data of patients were collected, including: gender, age, time of first onset, time of medication, clinical symptoms, number of recurrence, EDSS score, serum and cerebrospinal fluid AQP 4-IgG titers, imaging results, rheumatic immunity-related autoimmune antibodies, comorbidities, related adverse drug reactions, etc. Ten healthy volunteers with physical examination in our hospital were selected as the healthy control (HC) group.Blood (5ml) was collected from peripheral veins of patients and healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

All patients with NMOSD met the international consensus diagnostic criteria for NMOSD published in 2015. Before medication, TPMT activity was normal.

Exclusion Criteria:

Patients with fever, infection, or patients with other autoimmune diseases, uncontrolled malignancies, and other chronic diseases were excluded.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
The concentrations of 6-TGN and 6-MMPN in NMOSD patients | 1 month
  The mean 6-TGN concentrations and 6-MMPN concentrations in 1 month after AZA treatment were tested by HPLC
The concentrations of 6-TGN and 6-MMPN in NMOSD patients | 6 months
  The mean 6-TGN concentrations and 6-MMPN concentrations in 6 months after AZA treatment were tested by HPLC.
The concentrations of 6-TGN and 6-MMPN in NMOSD patients | 12 months
  The mean 6-TGN concentrations and 6-MMPN concentrations in over 12 months after AZA treatment were tested by HPLC.
Serum levels of IL-6, NLRP3 and IL-18 in NMOSD patients and HC | 1 month
  The levels of IL-6, IL-18, and NLRP 3 inflammasome were measured in the enzyme-linked immunoassay kit.
Serum levels of IL-6, NLRP3 and IL-18 in NMOSD patients and HC | 6 months
  The levels of IL-6, IL-18, and NLRP 3 inflammasome were measured in the enzyme-linked immunoassay kit.
Serum levels of IL-6, NLRP3 and IL-18 in NMOSD patients and HC | 12 months
  The levels of IL-6, IL-18, and NLRP 3 inflammasome were measured in the enzyme-linked immunoassay kit.

CONTACTS AND LOCATIONS:
Overall Officials: Yulan Tang, Study Director — First Affiliated Hospital of Guangxi Medical University
Locations (1):
- Qingmeng Huang, Nanning, Guangxi, China